CLINICAL TRIAL: NCT06228937
Title: Typing of Gut Microbiota in Patients With Limb Lymphedema and Recurrent Lymphangitis, a Prospective Observational Study
Brief Title: Gut Microbiota in Patients With Limb Lymphedema and Recurrent Lymphangitis
Acronym: LymphFM
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6208
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Lymphedema; Microbiota
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: patients affected by limb lymphedema with recurrent soft tissue infections
  Interventions: Other: analysis of a sample of stool
- Group B: patients affected by limb lymphedema without recurrent soft tissue infections
  Interventions: Other: analysis of a sample of stool

INTERVENTIONS:
Other: analysis of a sample of stool — typing of the gut microbiota from a stool sample

SUMMARY:
Lymphedema is a chronic and progressive disease of the lymphatic vessels which affects about 300 million people worldwide. Patients may experience recurrent soft tissue infection of the limb affected by lymphedema, in terms of erysipelas, lymphangitis or cellulitis. No previous study has ever investigated the possible role of the gut microbiota in the genesis of acute infectious/inflammatory episodes in these patients. Our hypothesis is that lymphedema patients with recurrent soft tissue infections are characterized by pro-inflammatory changes in the microbiota.

ELIGIBILITY:
Inclusion Criteria (Group A):

* 18-85 years
* primary or secondary, upper or lower limb lymphedema, I-II-III stage ISL
* at least 3 episodes of soft tissue infection in an year, in the last 2 years
* consent to participate in the study

Inclusion Criteria (Group B):

* 18-85 years
* primary or secondary, upper or lower limb lymphedema, stage I-II-III (ISL)
* no episodes of soft tissue infection in the last 2 years
* consent to participate in the study

Exclusion Criteria:

* No compliance to perform limb compression and skin hygiene
* Antibiotic therapy in the last 15 days
* Diabetes mellitus
* Immunodeficiency
* Ongoing neoplastic pathology
* Taking immunosuppressive drugs
* Unavailability to follow-up for at least 24 months post-enrollment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective observational cohort study will be conducted on patients with limb lymphedema, clinical stage I, II and III according to the International Society of Lymphology (ISL), followed by the Plastic Surgery Unit of the University Polyclinic A. Gemelli IRCCS. According to the positive or negative history for recurrent soft tissue infectious episodes, patients will be divided into two homogeneous groups for demographic and clinical characteristics (Groups A and B).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-02-22 (Estimated); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
comparison alpha diversity | 60 months
  comparison alpha diversity of the gut microbiota in groups A and B

SECONDARY OUTCOMES:
comparison beta diversity | 60 months
  comparison beta diversity of the gut microbiota in groups A and B
evaluation of the microbiome differential abundance | 60 months
  evaluation of the microbiome differential abundance to identify taxa associated

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No